CLINICAL TRIAL: NCT01968499
Title: Associations of the Pharmacogenetic and Pharmacokinetic Factors With Clopidogrel Low Response and Clinical Outcome in Patients With Coronary Stent Implantation: a Registration Study
Brief Title: Pharmacogenetic and Pharmacokinetic Study of Clopidogrel
Acronym: PPSC
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Chunjian Li, Professor, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: 002; NNSFC/81170181 (Other Grant/Funding Number: NNSFC/81170181)
Record Dates: First submitted 2013-10-17; First posted 2013-10-24 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Coronary Artery Disease
Keywords: coronary stent implantation; clopidogrel low response
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — DNA samples of all recuited patients are collected and stored for future analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All recruited patients: Patients who receive stent implantation and aged >18 years.

SUMMARY:
This registration study aims to investigate the associations of the pharmacogenetic and pharmacokinetic factors with clopidogrel low response and clinical outcome in patients with coronary artery disease, and provide new pharmacogenetic and pharmacokinetic targets for the individualized anti-platelet treatment.

DETAILED DESCRIPTION:
Associations of the Pharmacogenetic and Pharmacokinetic Factors With Clopidogrel Low Response and Clinical Outcome in Patients With Coronary Stent Implantation: a Registration Study

Published data linking clopidogrel non-responsiveness to adverse ischaemic events lead to the suggestion that the magnitude of platelet inhibition by clopidogrel can be monitored and individually adjusted. This has been tested in randomised clinical trials (ARCTIC, GRAVITAS and TRIGGER-PCI), but despite reducing platelet reactivity, a strategy of therapy adjustment based on platelet function monitoring did not reduce the incidence of cardiac ischaemic events1, which indicates that most pharmacodynamical tests monitored anti-platelet treatment failed so far.

We accordingly performed this registration study to investigate whether the pharmacogenetic and pharmacokinetic factors are associated with clopidogrel low response as well as clinical outcome, and aimed to provide new targets for the individualized anti-platelet treatment.

Inclusion criteria:

1. Successively recruit all patients who receive stent implantation and take aspirin 100 mg and clopidogrel 75 mg once daily (7:00 a.m.) for more than 5 days.
2. Patient aged >18 years;
3. Signed inform consent.

Exclusion criteria:

1. intolerant with aspirin or clopidogrel treatment (e.g. allergic reactions or gastrointestinal bleeding);
2. taking medication that could interfere with the antiplatelet efficacy of clopidogrel (e.g. vitamin K antagonists, direct oral anticoagulants or nonsteroidal anti-inflammatory drugs);
3. with myelodysplastic syndrome or abnormal baseline platelet counts of < 80 × 10∧9/L or > 450 × 10∧9/L;
4. hemoglobin < 90g/L;
5. with a history of cerebral hemorrhage within 1 year;
6. in pregnancy.

Clinical data collection:

1. Patients basic characteristics.
2. Diagnosis and complicated diseases.
3. Medical treatment and interventional treatment.

Methods:

Blood samples are collected 5 days after the patients' taking clopidogrel to perform the genetic testing and determine the light transmittancy aggregation (LTA) and the serum levels of the parent clopidogrel, intermediate and active metabolites of clopidogrel. LTA is to re-determined 1 month after clopidogrel consumption. Clopidogrel low response is defined as the inhibition of platelet aggregation (IPA) in response to 5μM ADP is more than 40%. Clinical follow-up will be performed 1month, 6month, and 1year after the patients' included. Major adverse cardiovascular events (MACE) is set as death, non-fatal myocardial infarction (MI), ischemic stroke. Associations of the pharmacogenetic and pharmacokinetic factors with clopidogrel low response and clinical outcome will be analyzed.

Tests:

1. ADP-induced platelet aggregation: LTA in response to 5μM ADP.
2. Arachidonic acid (AA)-induced platelet aggregation: LTA in response to 1mM AA.
3. Simultaneous detection of clopidogrel, 2-oxo-clopidogrel and its thiol metabolite in human plasma by the high performance liquid chromatography-tandem mass spectrometry (HPLC-MS/MS) method.
4. GWAS scan or genotyping of ABCB1,CYP2C19, paraoxonase 1 (PON1), CYP3A5, P2RY12.

Sample size: We plan to recruit 1800 patients.

Clinical follow-up: 1 month, 6 month, and 1 year after the patients' included.

Major adverse cardiovascular events (MACE): Death, non-fatal MI, ischemic stroke.

Minor adverse cardiovascular events: Hospitalization, revascularization, stent thrombosis (ARC definition) and minor, moderate, and major bleeding (TIMI definition).

ELIGIBILITY:
Inclusion Criteria:

1. Successively recruit all patients who receive stent implantation and take aspirin 100 mg and clopidogrel 75 mg daily for more than 5 days.
2. Patient aged >18 years;
3. Signed inform consent.

Exclusion Criteria:

1. intolerant with aspirin or clopidogrel treatment (e.g. allergic reactions or gastrointestinal bleeding);
2. taking medication that could interfere with the antiplatelet efficacy of clopidogrel (e.g. vitamin K antagonists, direct oral anticoagulants or nonsteroidal anti-inflammatory drugs);
3. with myelodysplastic syndrome or abnormal baseline platelet counts of < 80 × 10∧9/L or > 450 × 10∧9/L;
4. hemoglobin < 90g/L;
5. with a history of cerebral hemorrhage within 1 year;
6. in pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who receive stent implantation and aged >18 years.
Sampling Method: Probability Sample
Enrollment: 1805 (Actual)
Dates: Start 2011-03; Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Risk ratio | 1 year after patients' being recruited
  Risk ratio of the genotypes on MACE.
Risk ratio | 1 year after patients' being recruited
  Risk ratio of the pharmacokinetic results on MACE.

SECONDARY OUTCOMES:
Risk ratio | 1 month after patients' being recruited
  Risk ratio of the genotypes on clopidogrel low response.
Risk ratio | 1 month after patients' being recruited
  Risk ratio of the pharmacokinetic results on clopidogrel low response.

OTHER OUTCOMES:
Risk ratio | 1 year after patients' being recruited
  Risk ratios of the genotypes and pharmacokinetic results on the minor adverse cardiovascular events.

CONTACTS AND LOCATIONS:
Overall Officials: Chunjian Li, Ph.D, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Siller-Matula JM, Jilma B. Why have studies of tailored anti-platelet therapy failed so far? Thromb Haemost. 2013 Oct;110(4):628-31. doi: 10.1160/TH13-03-0250. Epub 2013 Jul 25. PMID 23884166
- [Derived] Zong J, Tang Y, Wang T, Ullah I, Xu K, Wang J, Chen P, Chen Z, Zhu T, Chen J, Li J, Wang F, Yang L, Fan Y, Shi L, Gong X, Eikelboom JW, Zhao Y, Li C. Impact of Insulin Receptor Substrate-1 rs956115 and CYP2C19 rs4244285 Genotypes on Clinical Outcome of Patients Undergoing Percutaneous Coronary Intervention. J Am Heart Assoc. 2022 Aug 16;11(16):e025058. doi: 10.1161/JAHA.121.025058. Epub 2022 Aug 5. PMID 35929455
- [Derived] Wang J, Wang J, Dong Z, Ma J, Teng J, Wang T, Zhang X, Gu Q, Ye Z, Ullah I, Tan C, Abdus S, Shi L, Gong X, Li C. An optimal window of platelet reactivity by LTA assay for patients undergoing percutaneous coronary intervention. Thromb J. 2021 Oct 19;19(1):73. doi: 10.1186/s12959-021-00323-5. PMID 34666778
- [Derived] Xu K, Ye S, Zhang S, Yang M, Zhu T, Kong D, Chen J, Xu L, Li J, Zhu H, Wang F, Yang L, Zhang J, Fan Y, Ying L, Hu X, Zhang X, Chan NC, Li C. Impact of Platelet Endothelial Aggregation Receptor-1 Genotypes on Platelet Reactivity and Early Cardiovascular Outcomes in Patients Undergoing Percutaneous Coronary Intervention and Treated With Aspirin and Clopidogrel. Circ Cardiovasc Interv. 2019 May;12(5):e007019. doi: 10.1161/CIRCINTERVENTIONS.118.007019. PMID 31018667
- [Derived] Ying L, Wang F, Zhang J, Yang L, Gong X, Fan Y, Xu K, Li J, Lu Y, Mei L, Zhou Z, Li C. Impact of hepatitis B virus (HBV) infection on platelet response to clopidogrel in patients undergoing coronary stent implantation. Thromb Res. 2018 Jul;167:119-124. doi: 10.1016/j.thromres.2018.04.017. Epub 2018 Apr 19. PMID 29807287